CLINICAL TRIAL: NCT04194502
Title: Intraoperative Coronary Artery Flow Patterns in Patients With Congenital Heart Disease and the Relationship to Short Term Surgical Outcomes.
Brief Title: Coronary Artery Assessement by TEE in Congenital Heart Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Lynne Nield, Staff Cardiologist, The Hospital for Sick Children
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 1000056046
Record Dates: First submitted 2019-11-12; First posted 2019-12-11 (Actual); Last update posted 2019-12-11 (Actual); Status verified 2019-12

CONDITIONS: Congenital Heart Disease
Keywords: Transesophageal echocardiography
MeSH Terms: conditions — Heart Defects, Congenital | interventions — Echocardiography, Transesophageal

STUDY DESIGN:
Intervention Model Description: The purpose of the study is to establish normal coronary artery pulse Doppler flow patterns and velocities using transoesophageal echocardiography (TEE) in patients with a variety of congenital heart disease
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pre-operative and intra-operative TEE (Other): All patients enrolled in the study will undergo a pre-op research TEE and a intra-op clinical transesophageal echo.
  Interventions: Diagnostic Test: Transesophageal echocardiogram (TEE)

INTERVENTIONS:
Diagnostic Test: Transesophageal echocardiogram (TEE) — All patients enrolled in the study will undergo a pre-operative research TEE and an intra-operative clinical TEE.

SUMMARY:
This study aims to establish normal coronary artery pulse Doppler flow patterns and velocities using transoesophageal echocardiography (TEE) in patients with a variety of congenital heart disease. This will be accomplished by performing pre-operative and intra-operative TEEs on up to 250 patients undergoing surgery for congenital heart disease.

DETAILED DESCRIPTION:
Little is known about coronary artery flow patterns in children. Invasive and non invasive studies in normal children have demonstrated that coronary artery flow velocities decrease with age and therefore heart rate. 'Normal' flow velocities in the left coronary artery are usually accepted between 0.3-0.6m/sec depending on age of the patient. Less is known about coronary flow patterns and velocities in patients with congenital heart disease. In addition the effects of coronary artery bypass and altered loading conditions may affect coronary flow patterns and velocities and in theory alter short and long term outcomes. This study hopes to is to establish normal coronary artery pulse Doppler flow patterns and velocities using transoesophageal echocardiography (TEE) in patients with a variety of congenital heart disease.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing surgical repair of congenital heart lesions at the Hospital for Sick Children between May 2017 and May 2018.

Exclusion Criteria:

1. Patients with hypoplastic left heart syndrome undergoing Norwood operation or Hybrid procedure
2. Patients who have undergone heart transplantation.
3. Patients were transoespphageal echocardiography is contraindicated (less than 3kg, recent upper gastrointestinal surgery).
4. Operations where TEE is not routinely indicated (patent ductus arteriosus ligation, aortic coarctation repair via a thoracotomy, vascular ring ligations).
5. Patients whose primary reason for surgery is coronary artery stenosis

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 118 (Actual)
Dates: Start 2017-04-19 (Actual); Primary Completion 2018-06-18 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
Coronary artery pulse doppler flow patterns will be assessed as normal or abnormal in patients with congenital heart disease | 5-7 minutes per TEE
  Pulse Doppler flow patterns in the LMCA, LAD, circumflex and RCA will be assessed as normal or abnormal using transoesophageal echocardiography (TEE) in patients with a variety of congenital heart disease
Measure the coronary artery pulse doppler flow velocities (cm/sec) in patients with congenital heart disease | 5-7 minutes per TEE
  The coronary artery pulse Doppler diastolic and systolic flow velocities (cm/sec) of the LMCA, LAD, circumflex and RCA will be assessed using TEE in patients with a variety of congenital heart disease.
Correlate pre-operative and post-operative coronary artery flow patterns abnormal and velocities (cm/sec) with negative post-operative clinical outcomes | Post-operative events will be collected from the time of discharge from the operating room until the participant is discharged from the hospital (typically between 3-14 days)
  Determine if there is a relationship between abnormal coronary artery flow patterns and velocities with negative post-operative clinical outcomes including death, delayed sternal closure, ECMO, ST segment changes, ventricular fibrillation or tachycardia, need for catheterization and stroke.

CONTACTS AND LOCATIONS:
Overall Officials: Lynne Nield, MD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No